CLINICAL TRIAL: NCT04751097
Title: The Intelligent Community Active Rehab for the Elderly Study Feasibility Study
Brief Title: The iCARE Feasibility Study
Acronym: iCARE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CUSH Health Ltd. (Industry)
Collaborators: University of Sussex (Other)
Responsible Party: Principal Investigator, Kalon Hewage, MBBS BSc MSc MRCS, Director and Co-Founder Cush Health, Trauma and Orthopaedic Registrar, CUSH Health Ltd.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: bsms9kd3
Record Dates: First submitted 2020-10-23; First posted 2021-02-11 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Accidental Fall
Keywords: feasibility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Platform (Experimental)
  Interventions: Other: CUSH Health Digital platform
- Routine Care (No Intervention)

INTERVENTIONS:
Other: CUSH Health Digital platform — Remote mobility monitoring and physiotherapy video app
  Arms: Digital Platform

SUMMARY:
Conducting assessment lower limb muscle strength, power and joint range of movement as well as inertial measurement unit (IMU) data capture during periods of walking and activities of daily living (sit to stand, stand to sit, climbing stairs) in participants over the age of 65. Assessing to see if there is any correlation between prospective follow up for incidence of fall events and patterns observed in the IMU data of the subject and to assess if the IMU data observed that results in higher or lower incidence of falls is related to any particular pattern in lower limb muscle strength, power and joint range of movement data.

DETAILED DESCRIPTION:
Research Question:

• What is the feasibility of conducting a large scale study to identify modifiable musculoskeletal factors, increasing the risk of falls in older adults; that can be detected in mobility data collected from a wearable device worn during activities of daily living?

Primary aim:

• To collect feasibility data on study processes, resource and management.

Secondary aims:

* Assess the preliminary efficacy of 'Wearable technology' in predicting falls risk in older adults during activities of daily living.
* Assess the preliminary efficacy of identifying musculoskeletal factors predisposing to mobility issues that are associated with or protective against falls.
* Assess the preliminary efficacy of specifically treating these musculoskeletal factors compared with traditional care?

ELIGIBILITY:
Inclusion Criteria:

* Aged over 65 years of age
* Able to give informed consent
* Able to mobilise independently or with mobility aid (walking stick, Zimmer frame etc.)

Exclusion Criteria:

* Patients under the age of 65.
* Patients who are bedbound or wheelchair bound.
* Patients with cognitive impairment and are unable to give informed consent.
* Significant medical co-morbidities that make participation in the study unsafe.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Total number of events fall at 1 week. | Recorded at day 7.
  Fall events are defined as an unintended action that leads to loss of balance or an unintended action that leads to unwanted movement towards the floor.
  This will be recorded as a numerical value of occurrence; For example if no fall events occur during the follow up period the the primary outcome measure will be reported as 0.
  Similarly if a participant has 4 fall events during the follow up period the primary outcome measure will be reported as 4.
  The minimum value will be 0 representing no fall events. Primary outcome values trending closer to 0 will be deemed a better outcome with 0 being the best.
  There is no defined maximum value but values trending away from 0 will be treated as a worse outcome.
Total number of events fall at 2 weeks. | Recorded at day 14.
  Fall events are defined as an unintended action that leads to loss of balance or an unintended action that leads to unwanted movement towards the floor.
  This will be recorded as a numerical value of occurrence; For example if no fall events occur during the follow up period the the primary outcome measure will be reported as 0.
  Similarly if a participant has 4 fall events during the follow up period the primary outcome measure will be reported as 4.
  The minimum value will be 0 representing no fall events. Primary outcome values trending closer to 0 will be deemed a better outcome with 0 being the best.
  There is no defined maximum value but values trending away from 0 will be treated as a worse outcome.
Total number of events fall at 1 month. | Recorded at day 30.
  Fall events are defined as an unintended action that leads to loss of balance or an unintended action that leads to unwanted movement towards the floor.
  This will be recorded as a numerical value of occurrence; For example if no fall events occur during the follow up period the the primary outcome measure will be reported as 0.
  Similarly if a participant has 4 fall events during the follow up period the primary outcome measure will be reported as 4.
  The minimum value will be 0 representing no fall events. Primary outcome values trending closer to 0 will be deemed a better outcome with 0 being the best.
  There is no defined maximum value but values trending away from 0 will be treated as a worse outcome.
Total number of events fall at 3 months. | Recorded at day 90.
  Fall events are defined as an unintended action that leads to loss of balance or an unintended action that leads to unwanted movement towards the floor.
  This will be recorded as a numerical value of occurrence; For example if no fall events occur during the follow up period the the primary outcome measure will be reported as 0.
  Similarly if a participant has 4 fall events during the follow up period the primary outcome measure will be reported as 4.
  The minimum value will be 0 representing no fall events. Primary outcome values trending closer to 0 will be deemed a better outcome with 0 being the best.
  There is no defined maximum value but values trending away from 0 will be treated as a worse outcome.
Total number of events fall at 6 months. | Recorded at day 180.
  Fall events are defined as an unintended action that leads to loss of balance or an unintended action that leads to unwanted movement towards the floor.
  This will be recorded as a numerical value of occurrence; For example if no fall events occur during the follow up period the the primary outcome measure will be reported as 0.
  Similarly if a participant has 4 fall events during the follow up period the primary outcome measure will be reported as 4.
  The minimum value will be 0 representing no fall events. Primary outcome values trending closer to 0 will be deemed a better outcome with 0 being the best.
  There is no defined maximum value but values trending away from 0 will be treated as a worse outcome.

SECONDARY OUTCOMES:
Timed up and go test (TUG test) | Completed at Day 1 and at the 6 months follow up.
  Total time taken for a participant to stand from a seated position walk forward 3 metres, turn around a marker, walk back towards the chair for 3 metres and sit back on the chair. Measured in seconds.
  A TUG test time of less than or equal to 13 seconds will be considered as a better outcome and a TUG test time of greater than 13 seconds will be considered a worse outcome.
Thirty second sit to stand test | Completed at Day 1 and at the 6 months follow up.
  Measured as the total number of repetitions of an activity (standing from a seated position then sitting down again) a participant is able to complete in 30 seconds.
  The minimum value is 0 which is a worse outcome and correlates with the participant unable to complete one repetition of the activity.
  There is no maximum value. Values of greater than or equal to 20 will be consider a better outcome.
2 min walk test | Completed at Day 1 and at the 6 months follow up.
  Total distance a participant is able to travel walking at a normal/ comfortable pace in 2 minutes. Measured in metres.
  The minimum value is 0 which is a worse outcome and correlates with the participant unable to move any distance within the allotted 2 minutes.
  There is no maximum value. Values of greater than or equal to 160 metres will be considered a better outcome.
Grip strength | Completed at Day 1 and at the 6 months follow up.
  The participant is asked to squeeze a dynamometer handle with one hand as hard as they can. The strength of their dominant and non-dominant hand measure independently. Measured in kilograms(Kg).
  The minimum value is 0 which is a worse outcome and correlates with the participant with no power.
  There is no maximum value. Values of greater than or equal to 20 will be consider a better outcome.
Timed stair climb | Completed at Day 1 and at the 6 months follow up.
  Power generated to climb stairs. Measured in Watts (W)
  This is calculated from:
  The height (vertical distance) of the stairs recorded in metres (m). The weight of the participant recorded in kilograms (kg). The time taken to climb the stairs recorded in seconds (s). The force of gravity set at 9.81
  Power = (weight x force of gravity x height of stairs) / time taken
Physical activity scale for the elderly (PASE) questionnaire | Completed at Day 1 and at the 6 months follow up.
  A brief (5 minutes) survey designed specifically to assess physical activity in studies of persons age 65 years and older. It combines information on leisure, household and occupational activity.
  It uses frequency, duration, and intensity level of activity over the previous week to assign a score, ranging from 0 to 793, with higher scores indicating greater physical activity thus a better outcome.
Short musculoskeletal function assessment (SMFA) questionnaire | Completed at Day 1 and at the 6 months follow up.
  The SMFA consists of two sections: (i) 34 questions cover- ing the assessment of the patients function and (ii) 12 questions covering how bothered patients are by their symptoms.The questionnaire is designed to be completed by the patient. It asks about patient experience over the previous week. Each question is scored 1 for no problems/no difficulty/ not bothered (depending on the question) to 5 for unable to do a task/symptoms all the time/being greatly bothered.
  The minimum value is 46 which is a better outcome. The maximum value is 230 which is a worse outcome.
Previous fall event history questions | Completed at Day1.
  Fall events are defined as an unintended action that leads to loss of balance or an unintended action that leads to unwanted movement towards the floor.
  This will be recorded as a numerical value of occurrence.
  Participants will be asked to answer how many fall events they have had prior to the start of the study:
  * In the last week
  * In the last month
  * In the last 3 months
  * In the last 6 months
  The minimum value will be 0 representing no fall events. Primary outcome values trending closer to 0 will be deemed a better outcome with 0 being the best.
  There is no defined maximum value but values trending away from 0 will be treated as a worse outcome.

IPD SHARING:
Plan to Share IPD: No